CLINICAL TRIAL: NCT00129636
Title: A Study to Determine the Usefulness of Patients Receiving Their Own Letter After an Outpatient Attendance Compared to Receiving a Copy of the Letter Being Sent to Their General Practitioner
Brief Title: The Usefulness of Patients Receiving Their Own Letter After an Outpatient Attendance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NHLICX3762
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Heart Diseases; Lung Diseases
Keywords: post consultation letter
MeSH Terms: conditions — Heart Diseases; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient attending hospital clinic (Other): patients were sent a letter especially dictated for them and a copy of the letter written by the hospital consultant to their GP to review
  Interventions: Procedure: Additional specific letter written to patient

INTERVENTIONS:
Procedure: Additional specific letter written to patient

SUMMARY:
As part of the NHS plan it has been proposed to extend some consultants' usual practices and to send all patients copies of the letters sent to their general practitioners (GPs) following outpatient consultations. The current Secretary of State for Health has further extended this proposal and suggested that patients should have a specific letter to themselves after a hospital consultation.

The aim of this study is to send patients both a copy of the letter sent to their GPs and a specific letter to themselves and to assess the usefulness and comprehensibility of each.

DETAILED DESCRIPTION:
As part of the NHS plan it has been proposed to extend some consultants' usual practices and to send all patients copies of the letters sent to their general practitioners following outpatient consultations. The current Secretary of State for Health has further extended this proposal and suggested that patients should have a specific letter to themselves after a hospital consultation.

The aim of this study is to send patients both a copy of the letter sent to their GPs and a specific letter to themselves and to assess the usefulness and comprehensibility of each. This study will assess the two styles of letter in Cardiology and Respiratory Outpatient Clinics staffed by 7 consultants and will involve a group of 15-20 patients from each of the clinics, total number approximately 150 patients.

All patients attending the clinics will be given a sheet outlining the study before their consultations. If they are interested in the study, patients will be given a Patient Information Sheet and asked consent to take part. The length of each of the two dictated letters will be recorded. To avoid costs to the NHS, the direct to patient letters will be typed at the study investigators' cost. Two copies of each letter, a short explanatory letter and a questionnaire will be sent to the patient and the patient will be asked to circle points in each of the letters which are unclear and return them to the department. At the end of the study the general practitioners will be contacted and asked their views about the two letters.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending respiratory/cardiology outpatient clinics

Exclusion Criteria:

* Patients with reading/language difficulties

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Comprehensibility of the two styles of letter | Baseline
  (length, reading ease, Flesch Kincaid Grade, items misunderstood)

SECONDARY OUTCOMES:
Patient preferences for the letters | baseline
  Patients indicated a preference for either the GP and patient letter or both
Deficiencies in the patient letter | baseline
  Deficiencies highlighted by the GP on the patient letter

CONTACTS AND LOCATIONS:
Overall Officials: Martyn R Partridge, MD FRCP, Principal Investigator — Imperial College London
Locations (1):
- NHLI Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roberts NJ, Partridge MR. How useful are post consultation letters to patients? BMC Med. 2006 Jan 20;4:2. doi: 10.1186/1741-7015-4-2. PMID 16426444